CLINICAL TRIAL: NCT01368523
Title: An Open-label, Multicenter Study of Oral AMN107 (Nilotinib) in Adult Patients With Imatinib - Resistant or - Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase Previously Enrolled to ENACT (CAMN107A2109) Trial
Brief Title: Study of Oral AMN107 (Nilotinib) in Adult Patients With Imatinib - Resistant or - Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase Previously Enrolled to CAMN107A2109 Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107APL01; EUDRACT 2008-000755-10 (Registry Identifier: EUDRACT)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Chronic Myelogenous Leukemia; chronic phase; accelerated phase; blastic phase; nilotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis | interventions — nilotinib

ARMS (1):
- nilotinib (Experimental)
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib
  Other Names: AMN107

SUMMARY:
The purpose of this study is to provide patients with imatinib resistant/intolerant chronic myeloid leukemia - in blast crisis, accelerated phase and chronic phase, who have been previously enrolled to CAMN107A2109 and benefit from the treatment, with access to nilotinib (AMN107) in Poland until such time as the treatment with this drug is financed by the National Health Found in Poland (via 'therapeutic program') or for a period of 18 months, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Imatinib - resistant or - intolerant Philadelphia chromosome-positive CML in chronic phase, accelerated phase or in blast crisis patients previously enrolled to CAMN107A2109 trial in Poland and continuing the treatment with nilotinib at the time of enrollment for this trial.
2. In the opinion of the investigators would benefit from the further treatment with nilotinib
3. No evidence of extramedullary leukaemic involvement, with the exception of liver and spleen
4. Males or females ≥18 years of age
5. WHO Performance Status of ≤ 2
6. QTc ≤ 450 msec on the average of three serial baseline ECG (using the QTcF formula).
7. Patients must have the following laboratory values:

   * Potassium within normal limits or corrected to within normal limits with supplements prior to the first dose of study medication
   * Total calcium (corrected for serum albumin) within normal limits or correctable with supplements
   * Magnesium within normal limits or corrected to within normal limits with supplements prior to the first dose of study medication
   * Phosphorus ≥ LLN or correctable with supplements
   * ALT and AST ≤ 2.5 x ULN or ≤ 5.0 x ULN if considered due to tumour
   * Alkaline phosphatase ≤ 2.5 x ULN unless considered due to tumour
   * Serum bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min
   * Serum amylase ≤ 1.5 x ULN and serum lipase ≤ 1.5 x ULN
8. Written signed and dated informed consent prior to any study procedures being performed.

Exclusion Criteria:

1. Known T315I mutations
2. Impaired cardiac function including any one of the following:

   * LVEF < 45% or below the institutional lower limit of the normal range (whichever is higher) as determined by echocardiogram
   * Inability to determine the QT interval on ECG
   * Complete left bundle branch block
   * Use of a ventricular-paced pacemaker
   * Congenital long QT syndrome or a known family history of long QT syndrome
   * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting brachycardia (< 50 beats per minute)
   * QTc > 450 msec on the average of three serial baseline ECG (using the QTcF formula). If QTcF > 450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc.
   * History of clinically documented myocardial infarction
   * History of unstable angina (during the last 12 months)
   * Other clinically significant heart disease (e.g. congestive heart failure or uncontrolled hypertension).
3. Known cytopathologically confirmed CNS infiltration (in absence of suspicion of CNS involvement, lumbar puncture not required)
4. Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection)
5. History of significant congenital or acquired bleeding disorder unrelated to cancer
6. Previous radiotherapy to ≥ 25% of the bone marrow
7. Major surgery within 4 weeks prior to Day 1 of study or who have not recovered from prior surgery
8. History of non-compliance to medical regimens or inability to grant consent
9. Use of therapeutic coumarin derivatives (i.e., warfarin, acenocoumarol, phenprocoumon)
10. Patients actively receiving therapy with strong CYP3A4 inhibitors (e.g, erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil) and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug or who are within 5 half-lives of the last dose of this medication prior to starting study drug.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
hematologic response | 18 months

SECONDARY OUTCOMES:
cytogenetic response | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Poland (3):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw